CLINICAL TRIAL: NCT07157514
Title: An Adaptive, Operationally Seamless Phase II / III Study of 131I-apamistamab-Led Allogeneic Hematopoietic Stem Cell Transplant in Patients With Relapsed or Refractory Acute Myeloid Leukemia With Active Disease
Brief Title: Radioimmunotherapy Conditioning With 131I- Apamistamab for Allogeneic Transplant in Relapse/Refractory AML
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIM-300
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Acute Leukemia; Myeloid Leukemia; Acute Myelogenous Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse; Myelogenous Leukemia; Myelogenous Leukemia, Acute; Myelogenous Leukemia in Relapse; Transplant-Related Disorder; Allogeneic Disease; Refractory AML
Keywords: Acute Myeloid Leukemia; Leukemia; Acute Myeloid; Acute Bone Marrow Cell Transplant; Transplant; Bone Marrow HCT; Refractory AML; Relapsed AML; I-131; Iomab; I131- Apamistamab; Iodine; Iodine-131; 131-I AML; Iomab-B; Radioimmunotherapy; Allogeneic Transplant; Radiotherapy; CD45; Anti-CD45 antibody; Apamistamab; Fludarabine; Bone Marrow Transplant; Radiolabeled antibody therapy; 131I -apamistamab
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute; Leukemia | interventions — fludarabine; Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: Adaptive, seamless Phase 2/3 design including Phase 2 randomized dose optimization followed by a Phase 3 randomized, controlled two-arm comparison of 131I-apamistamab conditioning versus control regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Experimental: I131-apamistamab + Fludarabine + TBI (Experimental): Participants receive a dosimetric dose and then a treatment dose of I131-apamistamab (at the marrow dose selected in Phase 2), followed by fludarabine 30 mg/m² IV daily on Days -6 through -2 and total body irradiation (TBI) 200 cGy on Day -1 prior to allogeneic hematopoietic stem cell transplant (HSCT) on Day 0.
  Graft-versus-host disease (GvHD) prophylaxis per investigator's choice:
  * Post-transplant cyclophosphamide (50 mg/kg on Days +3 and +4) + tacrolimus + mycophenolate mofetil, OR
  * Low-dose methotrexate + tacrolimus.
  Interventions: Drug: 131I-apamistamab; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation (TBI); Biological: Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
- Arm B: Active Comparator - Standard of Care Conditioning Regimen (Active Comparator): Participants receive standard of care conditioning regimen prior to allogeneic hematopoietic stem cell transplant (HSCT) on Day 0
  GvHD prophylaxis per investigator's choice:
  * Post-transplant cyclophosphamide (50 mg/kg on Days +3 and +4) + tacrolimus + mycophenolate mofetil, OR
  * Low-dose methotrexate + tacrolimus.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Allogeneic Hematopoietic Stem Cell Transplant (HSCT)

INTERVENTIONS:
Drug: 131I-apamistamab — Iodine-131 radiolabeled anti-CD45 monoclonal antibody (apamistamab). Administered IV as a dosimetric dose followed by treatment dose.
  Arms: Arm A: Experimental: I131-apamistamab + Fludarabine + TBI
Drug: Fludarabine — Fludarabine phosphate, 30 mg/m² IV daily on Days -6 through -2.
Drug: Cyclophosphamide — Cyclophosphamide
Radiation: Total Body Irradiation (TBI) — TBI, 200 cGy on Day -1 prior to HSCT.
  Arms: Arm A: Experimental: I131-apamistamab + Fludarabine + TBI
Biological: Allogeneic Hematopoietic Stem Cell Transplant (HSCT) — Unmodified, G-CSF-mobilized donor stem cells infused on Day 0.

SUMMARY:
This is a multicenter, open-label study in people aged 18 and older with relapsed or refractory acute myeloid leukemia. It has two parts. In Phase 2, we are testing three radiation dose levels of 131I-apamistamab combined with fludarabine and low-dose whole-body radiation before stem cell transplant to find the safest and most effective dose. In Phase 3, patients will be randomly assigned to receive either this treatment combination or a standard of care regimen before transplant. The main goal is to see if the new approach helps people live longer. Phase 2 will enroll about 60 people, and Phase 3 will enroll about 246 people.

DETAILED DESCRIPTION:
This trial consists of a Phase 2 randomized dose optimization component and a Phase 3 randomized, controlled two-arm component. This is a multicenter, open-label, study of 131I-apamistamab, fludarabine and TBI, which will be compared to standard of care regimen prior to HSCT in the Phase 3 portion, in subjects, aged 18 years old or greater, with active, relapsed or refractory AML. Active, relapsed or refractory AML is defined as any one of the following: (1) primary induction failure (PIF) after 2 or more cycles of therapy, or (2) first early relapse after a remission duration of fewer than 6 months, or (3) relapse refractory to salvage combination therapy, or (4) second or subsequent relapse.

All subjects will undergo screening prior to randomization in the study. Screening will include collection of informed consent, physical examination, review of inclusion/exclusion criteria with associated testing, summarizing documented history of AML and any other malignant disease, and identification and medical clearance of an appropriate allogeneic hematopoietic stem cell (HSC) donor.

Subjects must have active R/R AML with 5-20% blasts in marrow, documented CD45 expression, ≥18 years of age, not suitable for a myeloablative conditioning regimen, Karnofsky ≥70, and a medically cleared 8/8 matched HSC donor. Key exclusions include >20% marrow blasts, prior HSCT, prior maximal organ radiation, active CNS leukemia, significant cardiac disease, abnormal QTcF >450 ms, uncontrolled infection, or active malignancy within 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Have active, relapsed, or refractory AML with ≥5% and ≤20% blasts in the marrow.
2. 2R/R AML is defined as one of the following: Primary induction failure after ≥2 cycles of therapy, first early relapse after remission <6 months, relapse refractory to salvage combination therapy or second or subsequent relapse
3. Documented CD45 expression by leukemic cells via flow cytometry.
4. ≥18 years of age and not suitable for myeloablative conditioning regimen.
5. Circulating blast count <10,000/mm³ (hydroxyurea allowed).
6. Calculated creatinine clearance (Cockcroft-Gault) >50 mL/min.
7. Adequate hepatic function: AST/ALT ≤2 × ULN; total bilirubin ≤1.5 × ULN (≤3 × ULN if due to underlying malignancy or Gilbert's).
8. Karnofsky performance score ≥70.
9. Expected survival >60 days.
10. Central venous catheter line in place before study treatment.
11. 8/8 HLA-matched related or unrelated donor (HLA-A, HLA-B, HLA-C, DRB1).
12. Women of childbearing potential must be surgically sterile or use acceptable contraception through 1-year post-transplant.
13. Men with partners of childbearing potential must be surgically sterile or use acceptable contraception through 12 weeks after last dose.
14. Able to understand procedures, provide informed consent, and comply with study requirements.

Exclusion Criteria:

1. Positive human anti-mouse antibody (HAMA) at screening.
2. >20% leukemic blasts in marrow.
3. Prior radiation to maximally tolerated levels of any critical organ.
4. Active CNS leukemia (blasts in CSF or CNS chloromas).
5. Prior allogeneic or autologous HSCT.
6. Candidates suitable for myeloablative conditioning.
7. Clinically significant cardiac disease, including: NYHA Class III or IV heart failure, Clinically significant arrhythmias (ventricular tachycardia, ventricular fibrillation, Torsade de Pointes), Myocardial infarction with uncontrolled angina within 6 months, Clinically significant congestive heart failure or cardiomyopathy
8. QTcF >450 ms after correction of electrolytes (unless paced rhythm or investigator deems eligible; cardiology consult optional).
9. Positive HIV, HBV, or HCV test (exceptions: vaccinated HBV, or positive hepatitis markers with adequate organ function).
10. Active, uncontrolled infection.
11. Acute promyelocytic leukemia (t[15;17]).
12. Active malignancy within 2 years, except: Myelodysplastic syndrome, Treated non-melanoma skin cancer, Completely resected stage 0-1 melanoma (>1 year from resection), Carcinoma in situ or cervical intraepithelial neoplasia, Organ-confined prostate cancer without progression
13. Inability to tolerate diagnostic or therapeutic procedures, particularly radiation isolation.
14. Received anti-leukemic therapy within 14 days prior to randomization (hydroxyurea allowed up to day of 131I-apamistamab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) -Phase 3 | Up to 5 years post-randomization
  Defined as time from randomization to death from any cause. Subjects without documented death at the time of analysis will be censored at the date of last known contact.
Complete Remission (CR) at Day 28 Post-HSCT - Phase 2 | Day 28 post-HSCT
  Number of subjects achieving CR by Day 28 (±3 days) post-HSCT, based on bone marrow assessment.
Incidence of Grade ≥4 Non-Hematologic Toxicity | Up to 6 months post-HSCT
  Number and proportion of subjects developing grade ≥4 non-hematologic toxicities as graded by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Up to 5 years post-randomization
  Time from randomization to relapse, treatment failure, or death from any cause, whichever occurs first.
Relapse-Free Survival (RFS) | 6 months post-HSCT and up to 5 years post-randomization
  Probability of being alive without previous relapse of disease among subjects who achieve a post-transplant CR or CRi.
Overall Response Rate (ORR) | Day 28 post-HSCT and up to 12 months
  Proportion of subjects achieving complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) following transplant
Duration of Remission (DOR) | Up to 5 years post-randomization
  Time from first documented CR or CRi until relapse or death from any cause.
GvHD-Free Relapse-Free Survival (GRFS) | Up to 5 years post-HSCT
  Composite endpoint defined as time from HSCT to first event of grade III-IV acute GvHD, chronic GvHD requiring systemic therapy, relapse, or death.
Survival Rate at One and Two Years Post-Transplant | 1 year and 2 years post-HSCT
  Proportion of subjects alive at one year and two years following HSCT.
Engraftment | Day 100 post-HSCT
  Number of subjects achieving ≥95% donor cell engraftment by Day 100 post-HSCT.
Time to Engraftment | Up to Day 100 post-HSCT
  Days from HSCT (Day 0) until subject reaches ≥95% donor cell engraftment.
Incidence of Acute and Chronic GvHD | 6 months post-HSCT
  Number and proportion of subjects developing acute or chronic GvHD, summarized by severity.
Relapse-Free Survival (RFS) | 6 months post-HSCT
  Probability of being alive without relapse at 180 days among subjects achieving CR/CRi.
Overall Survival | Up to 2 years post-enrollment
  Time from enrollment to death from any cause.

OTHER OUTCOMES:
Minimal Residual Disease (MRD) Negativity Rate | Up to 12 months post-HSCT
  Proportion of subjects achieving MRD negativity by multiparameter flow cytometry among those with CR/CRi.
Adverse Events Related to Study Treatment | Up to 5 years post-randomization
  Number and proportion of subjects of adverse events due to study treatment, summarized by severity.
Adverse Events of Special Interest | Up to 5 years post-randomization
  Number and proportion of subjects of adverse events of special interest, summarized by severity.
Rates of Engraftment and Graft Failure | Up to Day 100 post-HSCT
  Rate evaluation of number of subjects achieving ≥95% donor cell engraftment or graft failure by Day 100 post-HSCT
Non-Relapse Mortality (NRM) | Up to 5 years post-randomization
  Time to deaths without relapse/recurrence
QTc Interval Prolongation | Up to 12 months post-HSCT
  Extended duration of the QT interval on an electrocardiogram
Incidence of Renal and Hepatic Toxicity | Up to 12 months post-HSCT
  Number and proportion of subjects developing renal and hepatic toxicity, summarized by severity.